CLINICAL TRIAL: NCT03780725
Title: An Open Label Phase I PET Imaging Study to Investigate the Bio-distribution and Tumor Uptake of [89Zr]Zr-BI 754111 in Patients With Advanced Non-small Cell Lung Cancer and Head and Neck Squamous Cell Carcinoma Treated With BI 754111 in Combination With BI 754091
Brief Title: This Study Tests How BI 754111 is Distributed in Patients With Advanced Non-small Cell Lung Cancer or Patients With Head and Neck Cancer Who Are Treated With BI 754091
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1381-0003; 2017-005046-30 (EudraCT Number)
Record Dates: First submitted 2018-11-26; First posted 2018-12-19 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial is divided in 2 Parts and will be conducted in a staggered approach, i.e. Part 2 follows Part 1. Part 2 will be initiated following a positive decision of the Study Monitoring Committee (SMC) after reviewing of all available data from Part 1 in order to assess whether a blockade of [89Zr]Zr-BI 754111 will be demonstrated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Ezabenlimab 240mg + BI 754111 600mg (Experimental)
  Interventions: Drug: BI 754111; Drug: [89Zr]Zr-BI 754111; Drug: BI 754091
- Part 2: Ezabenlimab 240mg + BI 754111 40mg (Experimental)
  Interventions: Drug: BI 754111; Drug: [89Zr]Zr-BI 754111; Drug: BI 754091

INTERVENTIONS:
Drug: BI 754111 — Solution for infusion
Drug: [89Zr]Zr-BI 754111 — Solution for infusion
Drug: BI 754091 — Solution for infusion
  Other Names: Ezabenlimab

SUMMARY:
The main objective of this study is to determine the biodistribution and intra-tumor accumulation of [89Zr]Zr-BI 754111 at baseline and its change upon treatment

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written Informed Consent Form (ICF) prior to any trial specific procedures, sampling, or analyses
* Patients of legal age (according to local legislation) at the time of signature of the ICF
* Patients with histologically confirmed diagnosis of recurrent NSCLC who received anti- PD-1 or anti PD-L1 as Part of last treatment with at least 3 months of stable disease (i.e.patients with confirmed response (PR or CR) regardless of duration of response or stable disease (SD) for a minimum of 3 months) and have become refractory to anti-PD- 1/ anti-PD-L1 based treatment OR

  --Patients with histologically confirmed diagnosis of recurrent metastatic HNSCC who progressed after platinum based therapy or not indicated for receiving standard (radio) chemotherapy (previous treatment with anti- PD-1/ PD-L1 is allowed)
* Eastern Cooperative Oncology Group (ECOG, R01-0787) score: 0 to 1
* Patient must have at least one PET imageable and evaluable tumor lesion of 20mm
* Patients must have at least one tumor lesion amenable to biopsy. This lesion should be PET imageable and evaluable as defined above and the biopsy should be obtained before first BI 754091 administration, unless medically contra-indicated. In the latter case, 25 4μm sections from an archival biopsy taken at relapse after the previous treatment are acceptable
* Must have evaluable lesion(s) according to Revised Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and iRECIST
* Life expectancy of at least 12 weeks after the start of the treatment according to the Investigator's judgement
* Male or female patients. Women of childbearing potential (WOCBP)1 and men able to father a child must be ready and able to use highly effective methods of birth control per International Conference on Harmonisation (ICH) M3 (R2) (that result in a low failure rate of less than 1% per year when used consistently and correctly) during trial Participation and for at least 6 months after the last administration of trial medication. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion Criteria:

* Not having fully recovered from major surgery before they enter into the trial according to investigator judgment or planned for major surgery within 12 months after screening, e.g. hip replacement
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled
* Previous treatment in this trial
* Any investigational or anti-tumor treatment within 4 weeks or within 5 half-life periods (whichever is shorter) prior to the initiation of trial treatment.
* Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 neuropathy due to prior platinum-based therapy
* Prior treatment with anti-LAG-3 agents
* Presence of other active invasive cancers other than the one treated in this trial, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment
* Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may Participate provided they are stable (i.e., without evidence of PD by imaging for at least 4 weeks prior to the first dose of trial treatment, and any neurologic symptoms have returned to baseline), and there is no evidence of new or enlarging brain metastases
* Inadequate organ function or bone marrow reserve as demonstrated by the laboratory values
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) >470 msec
  * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval
  * Ejection fraction <55% or the lower limit of normal of the institutional standard.
* History of pneumonitis within the last 5 years
* History of severe hypersensitivity reactions to other mAbs
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study treatment.
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy
* Active infection requiring systemic treatment (antibacterial, antiviral, or antifungal therapy) at start of treatment in this trial
* Known history of human immunodeficiency virus infection or an active hepatitis B or C virus infection
* Interstitial lung disease
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes him/her an unreliable trial patient or unlikely to complete the trial or unable to comply with the protocol procedures
* Women who are pregnant, nursing, or who plan to become pregnant in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC Locatie VUMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Miedema IHC, Huisman MC, Zwezerijnen GJC, Grempler R, Pitarch AP, Thiele A, Hesse R, Elgadi M, Peltzer A, Vugts DJ, van Dongen GAMS, de Gruijl TD, Menke-van der Houven van Oordt CW, Bahce I. 89Zr-immuno-PET using the anti-LAG-3 tracer [89Zr]Zr-BI 754111: demonstrating target specific binding in NSCLC and HNSCC. Eur J Nucl Med Mol Imaging. 2023 Jun;50(7):2068-2080. doi: 10.1007/s00259-023-06164-w. Epub 2023 Mar 2. PMID 36859619
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label Positron Emission Tomography (PET) imaging study to investigate the bio-distribution and tumor uptake of [89Zr]Zr-BI 754111 in patients with advanced non-small cell lung cancer and head and neck squamous cell carcinoma treated with BI 754111 in combination with BI 754091.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Part 1: Ezabenlimab 240mg + BI 754111 600mg: Baseline assessment phase (Cycle 1): 240 milligrams (mg) solution for infusion of BI 754091 (ezabenlimab) were administered by intravenous infusion on Day 1 of Cycle 1, followed by 4 milligrams solution for infusion of [89Zr]Zr-BI 754111 (4mg BI 754111 - 37 MBq) administered via intravenous infusion no later than Day 8 of Cycle 1.
  On-treatment phase (Cycle 2): 600 mg solution for infusion of BI 754111 together with 240 mg solution for infusion of BI 754091 (ezabenlimab) were administered by intravenous infusion on Day 1 of Cycle 2, followed by 4 milligrams solution for infusion of [89Zr]Zr-BI 754111 (4mg BI 754111 - 37 MBq) administered via intravenous infusion no later than Day 8 of Cycle 2.
  On-treatment phase (Cycle 3 and the following cycles): 600 mg solution for infusion of BI 754111 together with 240 mg solution for infusion of BI 754091 (ezabenlimab) were administered by intravenous infusion on Day 1 of each cycle.
  Each cycle last for 3 weeks. From Cycle 2 onwards, intravenous infusions of BI 754111 plus BI 754091 (ezabenlimab) once every 3 weeks until progression of disease, unacceptable toxicity, or maximum treatment duration of 1 year.
- Part 2: Ezabenlimab 240mg + BI 754111 40mg: Baseline assessment phase (Cycle 1): 240 milligrams (mg) solution for infusion of BI 754091 (ezabenlimab) were administered by intravenous infusion on Day 1 of Cycle 1, followed by 4 milligrams solution for infusion of [89Zr]Zr-BI 754111 (4mg BI 754111 - 37 MBq) administered via intravenous infusion no later than Day 8 of Cycle 1.
  On-treatment phase (Cycle 2): 40 mg solution for infusion of BI 754111 together with 240 mg solution for infusion of BI 754091 (ezabenlimab) were administered by intravenous infusion on Day 1 of Cycle 2, followed by 4 milligrams solution for infusion of [89Zr]Zr-BI 754111 (4mg BI 754111 - 37 MBq) administered via intravenous infusion no later than Day 8 of Cycle 2.
  On-treatment phase (Cycle 3 and the following cycles): 600 mg solution for infusion of BI 754111 together with 240 mg solution for infusion of BI 754091 (ezabenlimab) were administered by intravenous infusion on Day 1 of each cycle.
  Each cycle last for 3 weeks. From Cycle 2 onwards, intravenous infusions of BI 754111 plus BI 754091 (ezabenlimab) once every 3 weeks until progression of disease, unacceptable toxicity, or maximum treatment duration of 1 year.
Period: Overall Study
Arm/Group | Part 1: Ezabenlimab 240mg + BI 754111 600mg | Part 2: Ezabenlimab 240mg + BI 754111 40mg
Started | 3 | 5
Treated with at least one dose of Ezabenlimab and BI 754111 | 3 | 4
Completed | 0 | 0
Not Completed | 3 | 5
Not completed — Progression of disease | 3 | 4
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) : This patient set includes all patients who were documented to have received at least one dose of [89Zr]Zr-BI 754111, BI 754111, or BI 754091 (ezabenlimab).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Ezabenlimab 240mg + BI 754111 600mg | Part 2: Ezabenlimab 240mg + BI 754111 40mg | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (9.0) | 64.6 (8.6) | 64.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Standard Uptake Value (SUV) in a 1ml Sphere Around Highest SUV Pixel (SUVpeak) of [89Zr]Zr-BI 754111 for Tumor Uptake - Part 1
Description: The standardized uptake values (SUVs) are calculated as the ratios of the image derived radioactivity concentration upon the whole body concentration of the injected radioactivity, i.e. image derived radioactivity concentration / injected radioactivity concentration upon the whole body - a unitless value since the unit has been cancelled out. The Standard uptake value (SUV) in a 1 milliliter (mL) sphere around highest SUV pixel (SUVpeak) of [89Zr]Zr-BI 754111 for tumor uptake for part 1 participants is reported. The SUVpeak (also unitless since it is a SUV value) is summarized for each imaging time point (96hour, 144hour) as the mean tumor uptake over all selected lesions for each treatment cycle, respectively.
Time Frame: At 96 hours and 144 hours post-injection of [89Zr]Zr-BI 754111 in each cycle.
Population: Treated Set (TS): This patient set includes all patients who were documented to have received at least one dose of [89Zr]Zr-BI 754111, BI 754111, or BI 754091 (ezabenlimab). Only participants from part 1 are included in this analysis.
Measure: Mean (Standard Deviation); unit: SUV ratio
Arm/Group | Part 1: Ezabenlimab 240mg + BI 754111 600mg
Number analyzed (Participants) | 3
SUV ratio
  Cycle 1 (baseline phase) - 96 hours | 5.5 (1.0)
  Cycle 1 (baseline phase) - 144 hours | 5.2 (1.0)
  Cycle 2 (on-treatment phase) - 96 hours | 6.2 (2.7)
  Cycle 2 (on-treatment phase) - 144 hours | 7.0 (3.6)
Statistical Analysis 1: Comparison: Part 1: Ezabenlimab 240mg + BI 754111 600mg; The mean relative change is calculated as first deriving the relative change from baseline for each selected lesion at each time point (96hours, 144hours): 100 * (SUVpeak,lesion,timepoint,cycle2 - SUVpeak,lesion,timepoint,cycle1) / SUVpeak,lesion,timepoint,cycle1 Then, we calculate the mean over all evaluable lesions (at each time point) At last, the mean relative change is the lower mean value across time points; Test type: Other; Mean relative change from baseline = 17.1, Standard Deviation 47.7 — Mean relative change from baseline (Cycle 1) to on treatment (Cycle 2) is reported

2. Primary Outcome: Standard Uptake Value (SUV) in a 1ml Sphere Around Highest SUV Pixel (SUVpeak) of [89Zr]Zr-BI 754111 for Tumor Uptake - Part 2
Description: The standardized uptake values (SUVs) are calculated as the ratios of the image derived radioactivity concentration upon the whole body concentration of the injected radioactivity, i.e. image derived radioactivity concentration / injected radioactivity concentration upon the whole body - a unitless value since the unit has been cancelled out. The Standard uptake value (SUV) in a 1 milliliter (mL) sphere around highest SUV pixel (SUVpeak) of [89Zr]Zr-BI 754111 for tumor uptake for part 2 participants is reported. The SUVpeak (also unitless since it is a SUV value) is summarized for each imaging time point (96hour, 144hour) as the mean tumor uptake over all selected lesions for each treatment cycle, respectively.
Time Frame: At 96 hours and 144 hours post-injection of [89Zr]Zr-BI 754111 in each cycle.
Population: Treated Set (TS): This patient set includes all patients who were documented to have received at least one dose of [89Zr]Zr-BI 754111, BI 754111, or BI 754091 (ezabenlimab). Only participants from part 2 and have non-missing results are included in the analysis.
Measure: Mean (Standard Deviation); unit: SUV ratio
Arm/Group | Part 2: Ezabenlimab 240mg + BI 754111 40mg
Number analyzed (Participants) | 3
SUV ratio
  Cycle 1 (baseline phase) - 96 hours | 5.8 (4.4)
  Cycle 2 (on-treatment phase) - 96 hours | 4.6 (1.9)
  Cycle 1 (baseline phase) - 144 hours | 4.9 (3.6)
  Cycle 2 (on-treatment phase) - 144 hours | 4.3 (2.0)
Statistical Analysis 1: Comparison: Part 2: Ezabenlimab 240mg + BI 754111 40mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean relative change from baseline = -5.9, Standard Deviation 28.2 — Mean relative change from baseline (Cycle 1) to on treatment (Cycle 2) is reported

ADVERSE EVENTS:
Time Frame: From first dose of study medication until end of treatment + 30 days, up to 255 days.
Description: Treated Set (TS) : This patient set includes all patients who were documented to have received at least one dose of [89Zr]Zr-BI 754111, BI 754111, or BI 754091 (ezabenlimab).
Arm/Group | Part 1: Ezabenlimab 240mg + BI 754111 600mg | Part 2: Ezabenlimab 240mg + BI 754111 40mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ezabenlimab 240mg + BI 754111 600mg (N=3) | Part 2: Ezabenlimab 240mg + BI 754111 40mg (N=5)
Pyrexia (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Medical device site infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Device malfunction (Product issues) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ezabenlimab 240mg + BI 754111 600mg (N=3) | Part 2: Ezabenlimab 240mg + BI 754111 40mg (N=5)
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Candida infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Medical device site infection (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.

Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.

DOCUMENTS (2):
  • Study Protocol (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT03780725/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT03780725/SAP_001.pdf